CLINICAL TRIAL: NCT01663584
Title: Collection of Blood Samples for Development of Multi-disease Carrier Testing
Brief Title: Multi-disease Carrier Screening Test Validation
Status: Withdrawn | Type: Observational
Why Stopped: Samples were not needed for test development, therefore subjects were not recruited or enrolled
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Natera014
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Spinal Muscular Atrophy (SMA); Carrier Screening; Genetic Testing
Keywords: Spinal Muscular Atrophy (SMA); Carrier Screening; Genetic Testing
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Blood Specimen Collection

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — De-identified samples may be retained for future research.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood draw

SUMMARY:
The purpose of this study is to collect blood samples to enable validation of genetic testing for diseases within a multi-disease carrier screening panel. Samples will be collected from adult women or men who have previously tested positive as carriers for various recessive conditions. These are healthy adults who carry a mutation that might place them at increased risk of having a child with a specific genetic disorder. Study participation will be open to adults that were previously tested as part of their routine medical care and where test results demonstrated positive carrier status for a specific genetic disease. Samples will be tested for the disease mutation for which the subjects provides documentation of prior testing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Individuals who are carriers of an SMN1 deletion consistent with Spinal Muscular Atrophy carrier status and are able to provide documentation of carrier status determined from prior testing
* Able to provide a blood sample
* Pregnant women may be include in the study

Exclusion Criteria:

* Minors under the age of 18 years
* Individuals who are not carriers of a Spinal Muscular Atrophy mutation
* Individuals who are unable to provide documentation of Spinal Muscular Atrophy carrier status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participation will be open to individuals who have tested positive for carrier status of a specific genetic disease or mutation and are able to provide documentation of their test results.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Natera, Inc, San Carlos, California, United States